CLINICAL TRIAL: NCT05181774
Title: Prediction of Bleeding Risk After Anticoagulant Therapy for Atrial Fibrillation Based on Proteomics and Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yue LI (Other)
Responsible Party: Sponsor-Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: AF and stroke 2
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation; Bleeding; Anticoagulant Therapy
Keywords: Atrial Fibrillation; Bleeding; Anticoagulant therapy
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bleeding: After one-year follow-up, AF patients with anticoagulation-related bleeding complications were enrolled in this group.
  Interventions: Diagnostic Test: Proteomics; Diagnostic Test: Metabolomics
- Non-bleeding: After one-year follow-up, AF patients without anticoagulation-related bleeding complications were enrolled in this group.
  Interventions: Diagnostic Test: Proteomics; Diagnostic Test: Metabolomics

INTERVENTIONS:
Diagnostic Test: Proteomics — Proteomic data were obtained by LC-MS/MS Analysis-DIA platform.
Diagnostic Test: Metabolomics — Metabolomic data were obtained by UPLC-QTOF/MS platform.

SUMMARY:
Objectives: Atrial fibrillation (AF) is the most common arrhythmia. Anticoagulation with warfarin or new oral anticoagulants in patients with AF can significantly reduce thromboembolic events. However, due to the lack of bleeding risk predictors of oral anticoagulants, the bleeding risk of patients with AF cannot be accurately evaluated. The purpose of this study is to screen biomarkers that can predict bleeding in patients with AF through proteomics and metabolomics, and construct the protein metabolic network pathway of anticoagulant bleeding in patients with AF.

Design: AF patients treated with oral anticoagulants were enrolled in this study. Blood samples were centrifuged and the supernatant was stored in the refrigerator at - 80 ℃. All patients were followed up for one year to determine whether bleeding occurred after oral anticoagulants. Proteomic data were obtained by LC-MS/MS Analysis-DIA platform. Metabolomic data were obtained by UPLC-QTOF/MS platform. All of the omics data were used to compare proteins/enzymes with metabolic pathways. Quantitative changes of individual metabolites and proteins were calculated and graphed using the KEGG mapping tools.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Admission with atrial fibrillation or clinic visit for atrial fibrillation
3. Receive routine anticoagulant therapy;
4. Signing the consent form

Exclusion Criteria:

1. Pregnant women;
2. Lactating women;
3. Severe mitral stenosis;
4. Severe impairment of liver function;
5. Severe renal insufficiency;
6. Thyroid dysfunction requiring treatment;
7. Have a history of severe bleeding within five years, such as intracerebral hemorrhage and gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients treated with oral anticoagulants were enrolled in this study. Blood samples were centrifuged and the supernatant was stored in the refrigerator at - 80 ℃. All patients were followed up for one year to determine whether bleeding occurred after oral anticoagulants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers predicting bleeding in AF patients through proteomics and metabolomics. | 1 year
  Proteomic data were obtained by LC-MS/MS Analysis-DIA platform. Metabolomic data were obtained by UPLC-QTOF/MS platform.

SECONDARY OUTCOMES:
Protein metabolic network pathway of anticoagulant bleeding in patients with AF. | 1 year
  All of the omics data were used to compare proteins/enzymes with metabolic pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Yan, Harbin, Heilongjiang, China